CLINICAL TRIAL: NCT06853028
Title: The Role of Root Canal Treatment in Alleviating Endodontic Pain-Induced Asymmetry and Restoring Muscle Balance: a Prospective Cohort Study
Brief Title: The Role of Root Canal Treatment in Alleviating Endodontic Pain-Induced Asymmetry and Restoring Muscle Balance
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Kübra Gürler, DDS MSc, Cukurova University
Other Study IDs: 10.05.2024/144
Record Dates: First submitted 2025-02-14; First posted 2025-02-28 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Temporomandibular Disorders (TMD); Acute Apical Periodontitis of Pulpal Origin
Keywords: root canal treatment; ultrasonography; endodontic pain; acute apical periodontitis; masticatory laterality
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with a masticatory laterality due to acute apical periodontitis
  Interventions: Other: ultrasound measurement

INTERVENTIONS:
Other: ultrasound measurement — Muscle thickness measurements were performed with the ultrasound device immediately before root canal treatment, 1 week after, and 3 months after the treatment.

SUMMARY:
The study hypothesizes that masticatory laterality caused by acute apical periodontitis pain result in muscle asymmetry. Furthermore, it posits that successful root canal treatment, by restoring normal bilateral chewing function, will reduce this asymmetry, as evidenced by ultrasonographic measurements of the masseter and anterior temporal muscles.The main question it aims to answer is:

Can bilateral chewing function be restored after root canal treatment procedures in patients with masticatory laterality due to painful teeth due to acute apical periodontitis?

ELIGIBILITY:
Inclusion Criteria

* Patients with masticatory laterality due to tooth pain for at least 30 days
* First and second maxillary or mandibular molars with acute apical periodontitis due to deep caries
* Teeth with moderate or severe pain according to the VAS (no pain (0 mm), mild pain (1-3 mm), moderate pain (4-6 mm), and severe pain (7-10 mm))
* Teeth that responded positively to percussion test
* Teeth without periapical pathosis were included in the study. Exclusion Criteria
* Systemic conditions affecting muscle structure or function, such as neuromuscular or endocrine disorders.
* Non-endodontic odontogenic pain.
* Prior endodontic treatment of the relevant tooth within the last 30 days.
* History of trauma or surgery to the head, face, or teeth within the last six months.
* Severe communication disorders or psychological issues.
* Inability to complete treatment in a single visit due to exudation or bleeding
* Patients with masticatory laterality due to missing tooth on any side of the dental arch
* Patients who have painful teeth in opposite sides of the dental arch
* TMD patients were excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: •. 20 systemically healthy patients (11 female, 9 male) aged 18-60 years
  * Patients with masticatory laterality due to tooth pain for at least 30 days
  * First and second maxillary or mandibular molars with acute apical periodontitis due to deep caries
  * Teeth with moderate or severe pain according to the VAS (no pain (0 mm), mild pain (1-3 mm), moderate pain (4-6 mm), and severe pain (7-10 mm))
  * Teeth that responded positively to percussion test
  * Teeth without periapical pathosis
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Ultrasonography | immediately before root canal treatment, 1 week after and 3 months after the treatment
  Ultrasound (also called sonography or ultrasonography) is a noninvasive imaging test. An ultrasound picture is called a sonogram. Ultrasound uses high-frequency sound waves to create real-time pictures or video of internal organs or other soft tissues, such as blood vessels. The masseter and anterior temporal muscle thicknesses of the patients were measured bilaterally using a high-frequency linear scanning probe (7 MHz) in B-mode of the Clarius Mobile Health ultrasound device (Vancouver, Canada). As no established formula exists to calculate muscle thickness asymmetry, the asymmetry index was based on another study in the literature.
  Asymmetry Index = [(Control Side - Painful Side) / (Control Side + Painful Side)] × 100

CONTACTS AND LOCATIONS:
Locations (1):
- Çukurova Üniversitesi Diş Hekimliği Fakültesi, Gültepe, Sarıçam/Adana/Türkiye, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elbarbary M, Sgro A, Khazaei S, Goldberg M, Tenenbaum HC, Azarpazhooh A. The applications of ultrasound, and ultrasonography in dentistry: a scoping review of the literature. Clin Oral Investig. 2022 Mar;26(3):2299-2316. doi: 10.1007/s00784-021-04340-6. Epub 2022 Jan 14. PMID 35028733
- [Background] Jeon HM, Ahn YW, Jeong SH, Ok SM, Choi J, Lee JY, Joo JY, Kwon EY. Pattern analysis of patients with temporomandibular disorders resulting from unilateral mastication due to chronic periodontitis. J Periodontal Implant Sci. 2017 Aug;47(4):211-218. doi: 10.5051/jpis.2017.47.4.211. Epub 2017 Aug 21. PMID 28861285
- [Background] Daline IH, Slade GD, Fouad AF, Nixdorf DR, Tchivileva IE. Prevalence of painful temporomandibular disorders in endodontic patients with tooth pain. J Oral Rehabil. 2023 Jul;50(7):537-547. doi: 10.1111/joor.13457. Epub 2023 Apr 14. PMID 37021602
- [Derived] Gurler K, Guner Akgul I, Duyan Yuksel H, Sisli SN. The Role of Root Canal Treatment in Alleviating Endodontic Pain-Induced Asymmetry and Restoring Muscle Balance: A Self-Controlled Prospective Observational Study. Aust Endod J. 2025 Dec;51(3):650-659. doi: 10.1111/aej.12979. Epub 2025 Jul 29. PMID 40726276